CLINICAL TRIAL: NCT03930225
Title: Effectiveness of A Stigma Directed Interventional Program in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Noha Amer, Local Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MD/17.11.33
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Stigma, Social
Keywords: Stigma; Intervention program; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Social Stigma

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Outcomes Assessor
Masking Description: the outcome will be assessed by a different personnel than the investigator conducting the sessions of the intervention. The outcomes assessor will be blinded to which arm each participant belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): In the study group, both patients and their family members will be required to attend a weekly 1 hour long psycho-educational sessions. Moreover assessment sessions will be attended also.
  "The stigma directed intervention program"
  Interventions: Behavioral: Stigma Directed Psycho-educational Intervention program
- control group (Other): In the control group, only Patients will attend the psycho-educational sessions.
  Family members and patients will be required to attend the assessment sessions.
  Interventions: Behavioral: Stigma Directed Psycho-educational Intervention program

INTERVENTIONS:
Behavioral: Stigma Directed Psycho-educational Intervention program — psycho-educational intervention with emphasis on Stigma

SUMMARY:
randomized controlled study measuring the effectiveness of Stigma focused intervention in patients suffering from Schizophrenia

DETAILED DESCRIPTION:
Effectiveness of A Stigma Directed Intervention Program in Schizophrenia

It is a Randomized Controlled trial that aims at:

* Assessment of the relationship between self- stigma and

  1. Family burden on the caregiver (Family member).
  2. Medication adherence by patients.
* Assessment of the effectiveness of the family incorporation in the process of psychoeducation delivered to the patients suffering from Schizophrenia on the self-stigma and family burden of patients with Schizophrenia patients.

The study will be held in Mansoura University hospital Psychiatry department and will include 80 Egyptian patients with Schizophrenia or Schizoaffective disorder will be recruited from Psychiatry department of Mansoura University Hospital

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the diagnosis of schizophrenia or schizoaffective disorder according to DSM5.The clinical condition is stabilized.
2. Age range between 18 to 50 years.
3. Male and female sexes are included.
4. Availability of close relative in direct contact with the patient.

Inclusion Criteria for the family members:

1. Primary caregiver and the family member share household with patient.
2. No history of receiving treatment of psychiatric disorders.
3. No history of serious head trauma.

Exclusion Criteria :

1. Co morbid substance abuse or dependence disorder.
2. Co morbid intellectual disability.
3. Co morbid chronic medical or neurological condition or history of serious head trauma.

Exclusion Criteria for family members:

-Sever physical illness that hinders their participation- -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
change in Self-Stigma using the Arabic version of the internalized stigma of mental illness scale | Baseline assessment followed by Point 1 Assessment at the end of the 8 weekly sessions of the program ( after 2 months from baseline assessment) Final assessment after 3 months from point 1 Assessment
  stigma as experienced by patients themselves
change in perceived family burden using the perceived family burden scale | Baseline assessment---- followed by Point 1 Assessment at the end of the 8 weekly sessions of the program ( after 2 months from baseline assessment) Final assessment after 3 months from point 1 Assessment
  how much the disorder represent a burden on family
change in medication adherence using customized chart for each patient | Baseline assessment followed by Point 1 Assessment at the end of the 8 weekly sessions of the program ( after 2 months from baseline assessment) fFinal assessment after 3 months from point 1 Assessment
  the degree the patient adhere to the prescribed medications

SECONDARY OUTCOMES:
change in the clinical outcome using Positive and Negative Symptoms Scale | Baseline assessment followed by Point 1 Assessment at the end of the 8 weekly sessions of the program ( after 2 months from baseline assessment) Final assessment after 3 months from point 1 Assessment
  Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale. The scores for these scales are arrived at by summation of ratings across component items. Therefore, the potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. In addition to these measures, a Composite Scale is scored by subtracting the negative score from the positive score. This yields a bipolar index that ranges from -42 to +42, which is essentially a difference score reflecting the degree of predominance of one syndrome in relation to the other.

CONTACTS AND LOCATIONS:
Overall Officials: Vishwaijt Nimgaonkar, PhD, Study Chair — Pittsburgh university
Locations (1):
- Mansoura University Psychiatry Department, Al Mansurah, Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: No